CLINICAL TRIAL: NCT02764307
Title: Evaluation of Aerosol Delivery in Different Types of Nebulizers
Brief Title: Aerosol Delivery in Different Types of Nebulizers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Hui-Ling Lin, Assistant professor, Chang Gung University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ChangGungUniversity
Record Dates: First submitted 2016-04-25; First posted 2016-05-06 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aerosolized drug depositions (Experimental): Aerosol drug deposited on the inhaled and exhaled filters and the residual dose were evaluated delivered by four types of nebulizer: 1) a constant jet nebulizer, a breath enhanced nebulizer, a manual-actuated nebulizer, and a breath-actuated nebulizer.
  Interventions: Device: Constant jet nebulizer; Device: Breath enhanced nebulizer; Device: Manual-actuated nebulizer; Device: Breath-actuated nebulizer

INTERVENTIONS:
Device: Constant jet nebulizer — A constant jet nebulizer (Neb-easy, Galemed Corp., Taiwan) was tested with salbutamol sulfate powered by compressed gas flow at 6 L/min.
Device: Breath enhanced nebulizer — A breath enhanced nebulizer (Pari LC plus, Pari Inc., Germany) was tested with salbutamol sulfate powered by compressed gas flow at 6 L/min.
Device: Manual-actuated nebulizer — A manual-actuated nebulizer (A-T Neb, Atlantean Corporation, Taiwan) was tested with salbutamol sulfate powered by compressed gas flow at 6 L/min.
Device: Breath-actuated nebulizer — A breath-actuated nebulizer (AeroElipes, Trudell Medical Inc, Canada) was tested with salbutamol sulfate powered by compressed gas flow at 6 L/min.

SUMMARY:
Background: Nebulizers design influences efficiency of aerosol delivery. Performance of nebulizers is commonly tested by breathing simulators with static parameters. However, breathing patterns vary in adults.

Objectives: The purpose of this study was to evaluate drug deposition of different types of nebulizers testing with breathing patterns of healthy subjects.

DETAILED DESCRIPTION:
Material and Methods

The study was approved by Chang Gung Memorial Foundation Institutional Review Broad. Ten healthy subjects, aged 20.6±0.5 years, were recruited. Four nebulizers:

1. a constant jet nebulizer (Neb-easy, Galemed Corp., Taiwan);
2. a breath enhanced nebulizer (Pari LC plus, Pari Inc., Germany);
3. a manual-actuated nebulizer (A-T Neb, Atlantean Corporation, Taiwan); and
4. a breath-actuated nebulizer (AeroElipes, Trudell Medical Inc, Canada) were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy college subjects

Exclusion Criteria:

* Currently smoker
* History of asthma
* Drug allergy
* Pulmonary disease
* Heart disease
* Arrythmia
* Hyperthyroids
* Diabetes mellitus
* Lactacidosis
* Pregnant
* Under B-blocker medications

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Inhaled and exhaled drug concentrations | Drug deposition was tested Immediately after each nebulization, expected average of 20 minutes
  Drug deposited on the collecting filter was analyzed.

SECONDARY OUTCOMES:
Breathing parameters | During each nebulization testing, an expected average of 10 minutes
  Minute ventilation was recorded during nebulization

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Ling Lin, MSc, Principal Investigator — Chang Gung University

IPD SHARING:
Plan to Share IPD: Undecided